CLINICAL TRIAL: NCT01474564
Title: Feasibility of Obtaining and Characterizing Circulating Tumorigenic Cells in Patients With Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Adera Labs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-141
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Blood draw; pancreas; Tumorigenic Cells; 11-141
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Pts with Pancreatic Adenocarcinoma: This is an observational study to assess the feasibility of 1) isolating and enriching circulating tumorigenic cells from the peripheral blood of eligible pancreatic cancer patients and 2) successful gene expression profiling of these circulating tumorigenic cells.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Patients with pancreatic adenocarcinoma will be enrolled. Venous blood is collected in a standard 10 ml heparin blood collection tube. We may ask for blood samples at different times during the course of the study, specifically, before you start treatment and when your treatment changes. During the one year of the study, the physician anticipates blood samples will be collected a minimum of one and a maximum of four times. The amount of blood collected at any of these times will be 10 mL, about 1 tablespoon.

SUMMARY:
The purpose of this study is to collect blood samples and study cancer cells found in these blood samples from patients with pancreatic cancer. Prior research has discovered that tumor cells can be collected from the blood of patients with pancreatic and other cancers.

The physicians have developed techniques for isolating and analyzing cancer cells using a simple blood test. They will study how these cells relate to how chemotherapy works. They hope to use this information to guide choices of treatment for patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of pancreatic adenocarcinoma, confirmed at MSKCC.
* Patient eligible for chemotherapy treatment.
* Prior surgery, chemotherapy and/or radiation therapy for pancreatic adenocarcinoma is permitted.
* ECOG performance status 0-2.
* A minimum age of 18 years old.

Exclusion Criteria:

* Known to be HIV positive on antiretroviral therapy
* Prior organ allograft
* Any medical or psychiatric condition that may interfere with the ability to comply with protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
isolating and enriching circulating tumorigenic cells | 1 year
  A 10 mL blood sample will be drawn from participants prior to starting chemotherapy treatment. circulating tumorigenic cells from the peripheral blood of eligible pancreatic cancer patients. During the 1 year following enrollment, in the setting of disease progression, a subsequent 10 mL blood sample may be drawn from participants prior to changing chemotherapy treatment.

SECONDARY OUTCOMES:
successful gene expression profiling | 1 year
  of these circulating tumorigenic cells. For each blood sample collected, CTCs will be isolated, expanded, RNA extracted, gene expresion analysis performed and treatment profile sensitivity performed.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Yu, M.D., M.Sc., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/